CLINICAL TRIAL: NCT04080154
Title: A Single Arm, Open-label Study of Anlotinib in Patients With Hepatocellular Carcinoma (HCC) After Lenvatinib
Brief Title: Study of Anlotinib After Lenvatinib in Patients With Hepatocellular Carcinoma
Acronym: ALTER-H-002
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2019-173R
Record Dates: First submitted 2019-09-03; First posted 2019-09-06 (Actual); Last update posted 2020-04-03 (Actual); Status verified 2020-04

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — anlotinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anlotinib (Experimental): Anlotinib p.o., qd and it should be continued until disease progress or toxicity cannot be tolerated or patients withdraw consent.
  Interventions: Drug: Anlotinib

INTERVENTIONS:
Drug: Anlotinib — 12mg orally (p.o.) every day (qd) for 2 weeks of every 3 week cycle (i.e. 2 weeks on, 1 week off)

SUMMARY:
This clinical study evaluates the efficacy and safety of anlotinib in patients with hepatocellular carcinoma who have progressed on lenvatinib treatment. It is a single arm, open-label clinical trial conducted in China, and plan to recruit 28 patients. Primary endpoint of the study is Progress Free Survival.

DETAILED DESCRIPTION:
Anlotinib is a novel multi-target tyrosine kinase inhibitor (TKI) for tumor angiogenesis and proliferative signaling. The prime targets of anlotinib include receptor tyrosine kinases vascular endothelial growth factor receptor1 to 3 (VEGFR1-3), fibroblast growth factor receptor 1 to 4 (FGFR1-4), platelet-derived growth factor receptor α and β (PDGFR α, β), and stem cell factor receptor.

ELIGIBILITY:
Inclusion Criteria:

* Patients participate in the study voluntarily and sign informed consent.
* Histological or cytological confirmation of hepatocellular carcinoma (HCC) or non-invasive diagnosis of HCC as per Guidelines for Diagnosis and Treatment of Primary Liver Cancer in China (2017 Edition).
* Barcelona Clinic Liver Cancer stage Category C or B that cannot benefit from local treatment.
* Liver function status Child-Pugh Class A or Class B (≤7 points).
* Failure to prior treatment with lenvatinib according to the RECIST1.1. The last dose of lenvatinib should be over 2 weeks and within 10 weeks before the first dose of anlotinib.
* At least one measurable lesion according to the RECIST1.1.
* Eastern Cooperative Oncology Group Performance Status 0 or 1. Life expectancy of at least 3 months.
* Main organs function is normal. (normal main organs function as defined below: Hemoglobin (Hb) ≥ 90 g/L, Neutrophils (ANC) ≥ 1.5×109/L, Platelet count (PLT) ≥ 60×109/L, Albumin≥ 28g/L, Total bilirubin (TBIL) ≤ 2.0 × normal upper limit (ULN), Aspartate aminotransferase (AST) and Alanine aminotransferase (ALT) ≤ 3.0 ×ULN, Serum creatinine (Cr) ≤ 1.5× ULN, Hepatitis B virus DNA (HBV-DNA)<1000copy/ml.)
* The woman patients of childbearing age who must agree to take contraceptive methods (e.g. intrauterine device, contraceptive pill or condom) during the research and within another 6 months after it; who are not in the lactation period and examined as negative in blood serum test or urine pregnancy test within 7 days before the research; The man patients who must agree to take contraceptive methods during the research and within another 6 months after it.

Exclusion Criteria:

* Diagnosed with cholangiocellular carcinoma, mixed cell carcinoma and fibrolamellar hepatocellular carcinoma.
* History of other malignancy within 5 years or for now (except for non-melanoma skin cancer, cervix in situ carcinoma, superficial Bladder neoplasms).
* Liver function status Child-Pugh Class C, with malignant ascites.
* Any major unhealed wound, ulcer, or fracture occurred in a patient who had undergone major surgery or trauma within 4 weeks and/or had any bleeding or bleeding episodes which the degree is bigger than Common Terminology Criteria for Adverse Events (CTCAE) 3 grade within 4 weeks prior to enrollment.
* Participated in other anti-tumor clinical trials within 4 weeks.
* Prior systemic treatment for HCC, except lenvatinib. Intolerance of lenvatinib (defined as not less than 20 days at a minimum daily dose of 400 mg within the last 28 days).
* Symptoms that affect oral medication and cannot be controlled through proper treatment (such as inability to swallow, chronic diarrhoea and intestinal obstruction, etc.).
* Known history or symptomatic metastatic brain or meningeal tumors.
* Patients with arterial or venous thromboembolic events occurred within 6 months, such as cerebrovascular accident (including transient ischemic attack), deep vein thrombosis and pulmonary embolism.
* History of gastrointestinal bleeding due to severe gastroesophageal varices or definite tendency of gastrointestinal bleeding, or definite gastrointestinal bleeding tendency due to other causes, such as active ulcer, ulcerative colitis, etc. Fecal occult blood ≥ ++.
* Any of the following coagulation functions are abnormal, including: Prothrombin time (PT)>16 s, Activated partial thromboplastin time (APTT) >48 s, Thrombin time (TT)>21 s, International normalized ratio (INR)>2, fibrinogen (FIB)<2 g/L.
* Patients who underwent major surgery within 4 weeks.
* Patients who have got non remissive toxic reactions derived from lenvatinib treatment, which is over level 2 in CTC AE (4.0).
* Patients with any severe and/or unable to control diseases，including： Patients with unsatisfactory blood pressure control using antihypertensive drugs (systolic blood pressure ≥150 mmHg or diastolic blood pressure ≥100) mmHg); Patients with Grade 1 or higher myocardial ischemia, myocardial infarction or malignant arrhythmias(including QTc≥480ms) and patients with Grade 2 or higher congestive heart failure (NYHA Classification); Patients with active or unable to control serious infections, which is over level 2 in CTC AE (4.0); Patients with poorly controlled diabetes (fasting blood glucose(FBG)>10mmol/L); Patients with kidney failure who require hemodialysis or peritoneal dialysis; Patients with a history of immunodeficiency, including a positive HIV test or other acquired, congenital immunodeficiency disease, or a history of organ transplantation; Urine routine indicates that urine protein ≥ ++, and confirmed 24-hour urine protein quantitation > 1.0 g.
* Patients whose tumors had invaded important blood vessels by imaging or who, as determined by the researchers, were likely to invade important blood vessels during follow-up trial, resulting in fatal bleeding.
* Female patients who are pregnant or breastfeeding.
* Patients with drug abuse history and unable to get rid of or patients with mental disorders.
* Patients with concomitant diseases which could seriously endanger their own safety or could affect completion of the study according to investigators' judgment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2019-09-24 (Actual); Primary Completion 2021-02 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Progress free survival (PFS) | each 42 days up to progressive disease (PD) or death (up to 24 months)
  Progress free survival is defined as the time from first day of anlotinib treatment until the first date of either objective disease progression or death due to any cause, whichever occurs first.

SECONDARY OUTCOMES:
Overall Survival (OS) | From first day of anlotinib treatment until death (up to 24 months)
  Overall survival is defined as the time from first day of anlotinib treatment until the date of death due to any cause or the date of the last contact, at which the patients will be censored.
Objective Response Rate (ORR) | each 42 days up to intolerance the toxicity or PD (up to 24 months)
  Objective response rate is defined as the percentage of subjects whose best response was complete response (CR) or partial response (PR) according to the Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST1.1).
Disease Control Rate (DCR) | each 42 days up to intolerance the toxicity or PD (up to 24 months)
  Disease control rate is defined as the percentage of subjects whose best response was CR, PR or stable disease (SD) according to the RECIST1.1.
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | Until 30 day safety follow-up visit

CONTACTS AND LOCATIONS:
Overall Officials: Xiaowu Huang, doctor, Principal Investigator — Shanghai Zhongshan Hospital
Locations (1):
- 180 Fenglin Road, Shanghai, China